CLINICAL TRIAL: NCT07184840
Title: Eculizumab For Acute Attack of Neuromyelitis Optica Spectrum Disorder (NMOSD): a Multi-Center, Phase 2 Trial (EASE-NMO)
Brief Title: Eculizumab For the Acute Attack of Neuromyelitis Optica Spectrum Disorder
Acronym: EASE-NMO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Fu-Dong Shi, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2024-YX-456-01
Record Dates: First submitted 2025-09-08; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Neuromyelitis Optica Spectrum Disorder Attack
Keywords: Eculizumab; Acute Attack; Neuromyelitis Optica Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica | interventions — eculizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Methylprednisolone (IVMP) arm (Other): IVMP arm: 1000mg methylprednisolone x5d, oral prednisone 60mg, 5mg weekly decline + antibiotics
  Interventions: Drug: Intravenous Methylprednisolone (IVMP)
- IVMP+Eculizumab arm (Experimental): IVMP+Eculizumab arm: eculizumab (900 mg) will be administered intravenously once per week for a total of four doses (days 1, 8, 15, and 22) in conjunction with IVMP and oral prednisone (60mg, 5mg weekly decline).
  All enrolled patients will receive antibiotic prophylaxis against N meningitidis.
  Interventions: Drug: Intravenous Methylprednisolone (IVMP); Drug: Complement protein C5 inhibitor

INTERVENTIONS:
Drug: Intravenous Methylprednisolone (IVMP) — IVMP arm: 1000mg methylprednisolone x5d, oral prednisone 60mg, 5mg weekly decline + antibiotics
Drug: Complement protein C5 inhibitor — IVMP+Eculizumab arm: eculizumab (900 mg) will be administered intravenously once per week for a total of four doses (days 1, 8, 15, and 22) in conjunction with IVMP and oral prednisone (60mg, 5mg weekly decline).
  All enrolled patients will receive antibiotic prophylaxis against N meningitidis.
  Other Names: Eculizumab
  Arms: IVMP+Eculizumab arm

SUMMARY:
Neuromyelitis optica spectrum disorder (NMOSD) is a relapsing, inflammatory autoimmune disorder of the central nervous system characterized by the pathogenic anti-aquaporin 4 antibody (AQP4-IgG). The objectives of this study are to assess the efficacy and safety of eculizumab for treatment of patients with neuromyelitis optica spectrum disorders during acute phase who are anti-aquaporin-4 (AQP4) antibody-positive. Eculizumab, a humanized monoclonal antibody, inhibits the terminal complement protein C5 and prevents its cleavage into C5a and the formation of C5b-9 (MAC), has approved for preventive treatment of NMOSD. Given the high efficacy of C5 inhibition, eculizumab is proposed to potentially provide rapid relief from astrocyte destruction by reducing MAC formation, which could contribute to the fast alleviation of neurological deficit during NMO acute attack. The potential of eculizumab warrants further investigation as a treatment for acute neuromyelitis optica spectrum disorders attacks.

ELIGIBILITY:
Inclusion Criteria:

1. Anti-AQP4 antibody seropositive.
2. Male or female patients ≥18 years old
3. Body weight ≥ 35 kg
4. Acute optic neuritis and/or transverse myelitis enrolled within 28 days from the attack, with a change in neurological exam that meet an increase of OSIS at least 2 points of baseline compared to that of prior attack.
5. A female subject is eligible to enter the trial if she is:

   * Not pregnant or breastfeeding, not intending to conceive during the course of the trial

Exclusion Criteria:

1. Use of IVIg within 3 weeks prior to screening
2. Unresolved meningococcal infection
3. Any systemic bacterial or other infection which is clinically significant in the opinion of the Investigator and has not been treated with appropriate antibiotics
4. Participation in any other investigational drug study or was exposed to an investigational drug or device within 30 days of screening.
5. Has previously received treatment with eculizumab
6. Hypersensitivity to murine proteins or to one of the excipients of eculizumab
7. Any medical condition that, in the opinion of the Investigator, might interfere with thepatient's participation in the trial, poses any added risk for the patient, or confounds the assessment of the patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of improvement in OSIS from baseline to Day 28 by 2 points or more | Acute attack to Day 28
  The Optic-Spinal Impairment Score (OSIS) was developed to measure the disability status of subjects with demyelinating disease. It allows an objective quantification of the level of functioning that could be widely and reproducibly used by researchers and health care providers. OSIS score ranges from 0 to 25, which includes four primary functions: Visual Acuity (VA) (0-8), Motor Function (0-7), Sensory Function (0-5), and Sphincter Function (0-5). The higher scores reflect more severe disability. A decrease of at least 2 points in the overall OSIS score on day 28 compared to the baseline was regarded as a significant improvement.

SECONDARY OUTCOMES:
Change of OSIS from baseline to Day 28 | Acute attack to Day 28
  The Optic-Spinal Impairment Score (OSIS) was developed to measure the disability status of subjects with demyelinating disease. It allows an objective quantification of the level of functioning that could be widely and reproducibly used by researchers and health care providers. OSIS score ranges from 0 to 25, which includes four primary functions: Visual Acuity (VA) (0-8), Motor Function (0-7), Sensory Function (0-5), and Sphincter Function (0-5). Higher scores indicate more severe disability. A decrease in the overall OSIS score from baseline was used to measure neurological improvement.
Change of EDSS from baseline to Day 28 | Acute attack to Day 28
  EDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. EDSS consists of 7 FS (visual FS, brainstem FS, pyramidal FS, cerebellar FS, sensory FS, bowel and bladder FS, and cerebral FS) which are used to derive EDSS score ranging from 0 (normal neurological exam) to 10 (death from MS). A negative change from baseline in the overall EDSS score indicates neurological improvement.
Proportion of subjects that require plasma exchange or immunoadsorption at day 10 post treatment initiation. | Acute attack to Day 10
  PLEX Rescue was conducted only if a patient was not responding to the IVMP or IVMP+Eculizumab treatment as per the previous definition used; the assessment was made on day 10 after the IVMP/eculizumab initiation.
Change of OSIS from baseline to Day 7, 14, 21, and Week 12. | Acute attack to Week 12
  The Optic-Spinal Impairment Score (OSIS) was developed to measure the disability status of subjects with demyelinating disease. OSIS score ranges from 0 to 25, which includes four primary functions: Visual Acuity (VA) (0-8), Motor Function (0-7), Sensory Function (0-5), and Sphincter Function (0-5). A decrease in OSIS indicates improvement.
Change of EDSS from baseline to Day 7, 14, 21, and Week 12 | Acute attack to Week 12
  EDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. A decrease in EDSS indicates improvement.
Changes in Muscle Strength by MRC Scale for patients presenting with an acute relapse of myelitis at Days 7, 14, 21,28 and Week 12. | Acute attack to Week 12
  Muscle Power Assessment (MRC) was developed to assess the muscle power of limbs. A score of 0-5 was used to grade the power. Increasing disability of muscle power is reflected in an decreasing MRC score.
Changes in visual acuity in subjects presenting with an acute relapse of optic neuritis at Days 7, 14, 21,28, and Week 12 | Acute attack to Week 12
  Visual Acuity was measured with the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent of <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity.
Changes of pRNFL measured by OCT in subjects presenting with an acute relapse of optic neuritis at Days 28, and Week 12 | Acute attack to Week 12
  The peripapillary retinal nerve fiber layer (pRNFL) was analyzed by optical coherence tomography (OCT) measurements
Changes of mGCIPLT measured by OCT in subjects presenting with an acute relapse of optic neuritis at Day 28, and Week 12 | Acute attack to Week 12
  The macular ganglion cell-inner plexiform layer (mGCIPL) was analyzed by optical coherence tomography (OCT) measurements
To evaluate the changes of Nfl from baseline to Day 28 | Acute attack to Day 28
  Serum neurofilament light chain (NfL): Blood sample will be obtained to determine the level of Nfl.
To evaluate the changes of GFAP from baseline to Day 28 | Acute attack to Day 28
  Glial Fibrillary Acidic Protein (GFAP):Blood sample will be obtained to determine the level of GFAP.
To evaluate the changes of complement activity (CH50) from baseline to Day 28 | Acute attack to Day 28
  CH50: Blood sample will be obtained to determine the hemolytic activity of serum complement.
To compare the change in MRI lesion size by T2 weighted imaging and T1 post-contrast imaging from baseline to Week 12 | Acute attack to Week 12
  MRIs will be analyzed for counting the numbers of new lesions by T2 hyper-intensity in the brain, spinal cord and optic nerve, and the volume of T1 post-contrast enhancement.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No